CLINICAL TRIAL: NCT06522438
Title: Early Healing Dynamics and Microbial Changes Following the Use of a Novel Thermosensitive Gel With Hyaluronic Acid and Octenidine as an Adjunct to Non-surgical Periodontal Treatment
Brief Title: Hyaluronic Acid and Octenidine Gel as an Adjunct to Non-surgical Periodontal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 346806
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Periodontitis; Wound Heal; Periodontal Pocket; Periodontal Inflammation; Periodontal Attachment Loss
Keywords: Hyaluronic Acid; Octenidine; Biomarkers; Non-surgical periodontal treatment
MeSH Terms: conditions — Periodontitis; Periodontal Pocket; Periodontal Attachment Loss | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Non-surgical periodontal treatment (NSPT) plus Hyaluronic Acid (HA) and Octenidine gel.
  Interventions: Combination Product: Hyaluronic Acid (HA) and Octenidine gel; Procedure: Non-surgical periodontal treatment (NSPT)
- Control Group (Active Comparator): Non-surgical periodontal treatment (NSPT) alone.
  Interventions: Procedure: Non-surgical periodontal treatment (NSPT)

INTERVENTIONS:
Combination Product: Hyaluronic Acid (HA) and Octenidine gel — A thermosensitive gel with Hyaluronic Acid (HA) and Octenidine (Pocket-X®, Geistlich, Wolhusen, Switzerland) will be applied in the periodontal pockets ≥5mm immediately after the subgingival PMPR, by means of a pre-filled syringe bearing a thin plastic tip and following manufacturer's instructions.
  Arms: Test Group
Procedure: Non-surgical periodontal treatment (NSPT) — Full mouth supragingival professional mechanical plaque removal (PMPR) and subgingival PMPR at sites with PPD ≥4mm will be performed with the aid of manual and power-driven instruments under local anaesthesia.

SUMMARY:
This parallel-group, pilot study will test the hypothesis that the adjunctive use of a thermosensitive gel containing Hyaluronic Acid (HA) and Octenidine to non-surgical periodontal treatment (NSPT) will be able to modulate the early wound healing events. This will be assessed through the expression of specific gingival crevicular fluid markers, as well as by changes in gingival blood flow (assessed by laser speckle contrast imaging), bacterial load, soft tissues contour, clinical parameters and patient-reported outcomes.

The study will involve up to 26 patients and will take place at the Centre for Oral Clinical Research (COCR), at the Institute of Dentistry, Faculty of Medicine and Dentistry, Queen Mary University of London under The Royal London Dental Hospital, Barts Health NHS Trust. Patients will be randomised to receive either NSPT alone or NSPT+ HA and Octenidine gel, and will be followed up to 3 months after treatment.

The study will consist of 7- 8 visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and above
* Engaged patients presenting with a Full Mouth Plaque Score (FMPS) of ≤ 20% within the 6 weeks prior to enrolment, or exhibiting a ≥ 50% reduction in plaque score from the initial screening visit.
* Periodontitis stage III/IV (grades A to C) with at least one site per quadrant with PPD ≥5mm, bleeding on probing and attachment loss ≥5mm
* Willing to sign informed consent and comply with study procedures

Exclusion Criteria:

* Know hypersensitivity and/or allergy to any of the product's component (as per user leaflet)
* Self-reported pregnancy or lactation
* Smoking (current or in past 5 years), including e-cigarettes/vaping
* Medical history including diabetes mellitus or other serious medical/ psychiatric conditions or transmittable diseases that according to the investigator may increase the risk associated with study participation
* History of conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures or/and systemic antibiotic therapy during the 3 months preceding the baseline evaluation
* In chronic treatment with anti-inflammatory (including corticosteroids), anticoagulants/antiplatelets (including aspirin), immunosuppressants or other medication that can severely impact wound healing
* History of alcohol or drug abuse
* Subgingival professional mechanical plaque removal (excluding not-extensive subgingival debridement as judged by the examining clinician) and/or surgical periodontal treatment within the last 12 months
* Other severe acute or chronic medical or psychiatric condition or psychological disorder, including limited mental capacity or language skills such that study information could not be understood, informed consent could not be obtained, or simple instructions could not be followed, or any additional conditions which, in the judgement of the investigator, would make the subject inappropriate for entry into this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the expression of GCF wound healing biomarkers | Baseline, 1, 7, 15, 30 days and 3 months following treatment
  Changes in the expression of GCF wound healing biomarkers at 1, 7, 15, 30 days and 3 months following treatment will be assessed. A subset of analytes involved in the healing process and signalling pathways such as i) inflammation/immune response (e.g., IL-1 β, IL-1 α, IL-6, IL-8, IL-4, IL-10,IL-17, TNF- α, MMP-1, MMP-8, MMP-9, TIMP-1), ii) bone formation/resorption (e.g., TGF- β, osteocalcin, osteopontin, osteoprotegerin, BMP-2), iii) oxidative stress (e.g., Myeloperoxidase), and iv) angiogenesis (e.g., VEGF, angiopoietin-1) will be selected based on the pathways identified and optimized in the genomic and proteomic work from our group. Multiplex immunoassays will be designed specifically for quantitative analyses in the GCF for the 2 groups at the different time points.

SECONDARY OUTCOMES:
Changes in the Blood flow | Baseline and at 1, 7, 15, and 30 days following treatment.
  Changes in the blood flow at 1, 7, 15, and 30 days following treatment, evaluated with Laser Speckle Contrast Imaging (LSCI)
Changes in the bacterial load | Baseline and at 7, 15, 30 days and 3 months following treatment.
  Changes in the bacterial load associated with treated sites at 7, 15, 30 days, and 3 months following intervention. Subgingival plaque samples will be analysed using next generation marker DNA sequencing to characterise the subgingival microbiota to identify and determine the levels of key periodontal bacterial pathogens and microbial community-wide changes in sites treated at the different time points.
Changes in the probing pocket depth (PPD) | Baseline and at 3 months after intervention
  PPD will be measured in mm using a University of North Carolina (UNC-15) periodontal probe at six sites per tooth (i.e., mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual).
Changes in the gingival recession (REC) | Baseline and at 3 months after intervention
  REC will be measured in mm using a University of North Carolina (UNC-15) periodontal probe at six sites per tooth (i.e., mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual).
Changes in the clinical attachment level (CAL) | Baseline and at 3 months after intervention
  CAL will be calculated considering the values for PPD and REC in mm
Changes in the Full mouth plaque score (FMPS) | Baseline and at 3 months after intervention
  FMPS will be recorded as a percentage of total surfaces (6 sites per tooth), which reveal the presence of plaque. A binary score will be assigned to each surface (1 for plaque present, 0 for absent).
Changes in the Full mouth bleeding score (FMBS) | Baseline and at 3 months after intervention
  FMBS will be recorded as percentage of total surfaces (6 aspects per tooth/implant), which reveal the presence of bleeding within 10 - 30 seconds following periodontal probing. A binary score will be assigned to each surface (1 for bleeding present, 0 for bleeding absent).
Changes in the suppuration | Baseline and at 3 months after intervention
  Suppuration will be recorded as percentage of total surfaces (6 aspects per tooth), which reveal the presence of suppuration following periodontal probing. A binary score will be assigned to each surface (1 for suppuration present, 0 for suppuration absent).
Soft tissues contour changes | Baseline, 1, 7, 15, 30 days, and 3 months following treatment
  Soft tissues contour changes will be assessed at 1, 7, 15, 30 days, and 3 months following treatment. An intra-oral 3D scanner will be used to capture and monitor soft tissue contour changes during early phase of healing. The obtained images will be then superimposed (baseline and follow-ups) and calculation of linear and volumetric changes of the soft tissue (magnitude of the swelling, changes in shape and volume) will be performed.
Changes in the periodontal inflamed surface area (PISA) | Baseline and at 3 months after intervention
  The periodontal inflamed surface area (PISA) is expressed in mm2 and will be calculated as the sum of the PPD of BOP-positive sites for the total dentition, which can be easily calculated using routine periodontal charting.
Dentin hypersensitivity | Baseline, 1, 7, 15, 30 days, and 3 months after procedure
  A 100-mm horizontal visual analog scale (VAS) will be used to assess dentine hypersensitivity. The VAS is scored from 0= none to 100= worst dentin hypersensitivity possible and the subject will indicate the degree by marking vertically across the VAS scale.
Patient perception about therapy | 1,7 and 15 days after procedure
  The extent of discomfort and/or pain experienced will be evaluated using a 100-mm visual analog scale (VAS). The anchors for each end of the scales will be designated as 0=none to 100= worst. The extent of oedema, hematoma, high fever, and interference in daily activities during the initial weeks will also be evaluated in the same way.
Global changes in quality of life | 3 months after procedure
  Periodontal health and quality of life following periodontal therapy will be measured through specific questionnaire at 3 months after treatment. Questionnaire will include questions to evaluate patient's perception of treatment on their periodontal health and quality of life. Patients will answer by selecting one of the following options: worsened a lot, worsened a little, stayed the same, improved a little, improved a lot, or don't know.

CONTACTS AND LOCATIONS:
Overall Officials: Jeniffer Perussolo, DDS, MS, PhD, Principal Investigator — QMUL
Locations (2):
- United Kingdom (2):
  - Centre for Oral Clinical Research (COCR), London
  - The Royal London Dental Hospital, Barts Health NHS Trust, London